CLINICAL TRIAL: NCT01944540
Title: Comparison of Coventional Endoscopic Submucosal Dissection and Optimized Endoscopic Submucosal Dissection With Snaring for Colorectal Neoplasm
Brief Title: Brief Title : Optimized Endoscopic Submucosal Dissection With Snaring for Colorectal Neoplasm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Sik Byeon, Asan Medical Center, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: optESDs2013AMC
Record Dates: First submitted 2013-09-13; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional ESD (Active Comparator): Conventional ESD arm indicates the group in which conventional ESD method is applied for the dissection of colorectal neoplasm.
  Interventions: Procedure: Conventional ESD
- Optimized ESD with snaring (Experimental): Optimized ESD with snaring arm indicates the group in which optimized ESD with snaring method is applied for the dissection of colorectal neoplasm.
  Interventions: Procedure: Optimized ESD with snaring

INTERVENTIONS:
Procedure: Optimized ESD with snaring
  Arms: Optimized ESD with snaring
Procedure: Conventional ESD
  Arms: conventional ESD

SUMMARY:
This study is aimed to analyze the outcomes after conventional endoscopic submucosal dissection (ESD) and optimized ESD with snaring (oESD-S) for colorectal neoplasm that is more than 20 mm in diameter of laterllay spreading tumor or flat elevated lesion without stalk.

Optimized ESD with snaring means submucosal dissection followed by snaring when narrowed circumference of the remained submucosal tissue beneath the lesion is less than 5 mm in diameter with snaring, then resected by using an electric current.

The investigators expect optimized ESD with snaring can provide more time-saving procedure with comparable en-bloc resection rate and perforation rate, when compared with the conventional ESD method.

ELIGIBILITY:
Inclusion Criteria:

* colorectal laterally spreading tumor that is more than 20 mm in diameter
* other elevated or flat colorectal neoplasm without stalk, that is more than 20 mm in diameter

Exclusion Criteria:

* colorectal neoplasms that are proven or suspected to be invaded more than submucosal invasion
* colorectal neoplasms that have severe fibrosis beneath the target lesion
* patient's refusal to participate this study
* less than 18 years old
* subjects who cannot consent voluntarily due to the communication difficulty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
procedure time | 8 months
En Bloc resection rate | 8 months

SECONDARY OUTCOMES:
histologic complete resection rate | 8 months
complication rate | 8 months
  perforation rate, bleeding rate

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Sik Byoen, MD, Principal Investigator — Department of Gastroenterology, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Bae JH, Yang DH, Lee S, Soh JS, Lee S, Lee HS, Lee HJ, Park SH, Kim KJ, Ye BD, Myung SJ, Yang SK, Byeon JS. Optimized hybrid endoscopic submucosal dissection for colorectal tumors: a randomized controlled trial. Gastrointest Endosc. 2016 Mar;83(3):584-92. doi: 10.1016/j.gie.2015.06.057. Epub 2015 Aug 28. PMID 26320696